CLINICAL TRIAL: NCT01753297
Title: A Multicentric, Multinational (China and Russia), Randomised, Open, Controlled Study of Immediate 9 Months Adjuvant Hormone Therapy With Triptorelin 11.25 mg Versus Active Surveillance After Radical Prostatectomy in High Risk Prostate Cancer Patients
Brief Title: A Study of Immediate 9 Months Adjuvant Hormone Therapy With Triptorelin 11.25 mg Versus Active Surveillance After Radical Prostatectomy in High Risk Prostate Cancer Patients.
Acronym: PRIORITI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-38-52014-194
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triptorelin, 11.25 mg (Active Comparator): Triptorelin, powder and solvent for suspension (prolonged released form)
  Interventions: Drug: Triptorelin 11.25 mg
- Active surveillance (No Intervention): Active surveillance after radical prostatectomy (RP)

INTERVENTIONS:
Drug: Triptorelin 11.25 mg — Triptorelin, one injection every 3 months. A total of 3 injections (at baseline, 3 and 6 months)
  Arms: Triptorelin, 11.25 mg

SUMMARY:
The purpose of this study is to assess the benefit of immediate hormonal treatment after Radical Prostatectomy in Chinese and Russian patients with high risk prostate cancer. To reach this target, the trial will compare a group of patients treated with triptorelin at 8 weeks after the surgery and for a duration of 9 months (3 injections) versus another group (called "active surveillance group") who will be not receiving triptorelin. Both groups will be followed every 3 months to monitor any sign of disease progression during a minimum of 36 months

DETAILED DESCRIPTION:
This trial is a phase IV (in Russia and China) as approved indication is locally advanced or metastatic prostate cancer in both countries.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed adenocarcinoma of the prostate
* Radical Prostatectomy with curative intent performed no more than 8 weeks before randomisation
* High risk criteria of disease progression, defined as follows:

Gleason score ≥8 on prostatectomy specimen, and/or Pre RP PSA level ≥20 ng/mL, and/or Primary tumour stage 3a (pT3a) (with any PSA level and any Gleason score)

* Post-RP PSA levels ≤0.2 ng/mL at 6 weeks

Exclusion Criteria:

* Evidence of lymph nodes or distant metastasis
* Positive margins
* Evidence of any other malignant disease, not treated with a curative intent
* Had surgical castration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (18):
- China (9):
  - Chinese PLA General HospitalDepartment of UrologySite #156007, Beijing
  - Peiking University First Hospital Site #156011, Beijing
  - West China Hosspital, Sichuan UniversityDepartment of Urology Site #156008, Chengdu
  - The First Affiliated Hospital of the 3th Military Medical University of PLA (Southwest Hospital) Site # 156010, Chongqing
  - SUN YAT-SEN Cancer Center Department of Site #156009, Guangzhou
  - The third hospital affiliated to Sun Yat-sen University Site #156005, Guangzhou
  - The first hospital affiliated to medical school of Zhejiang university Site #156001, Hangzhou
  - Fudan University cancer hospital Site #156003, Shanghai
  - First Affiliated Hospital of the Fourth Military Medical University Site #156004, Xi'an
- Russia (9):
  - SIH Altaian Territorial Oncological Dispensary Site #643006, Barnaul
  - FSBI "Research Institute of Urology" of Ministry of health care of Russia Site #643002, Moscow
  - State Budgetary Healthcare Institution "Moscow Clinical Scientific-Practical Center named after A. S. Loginov of Healthcare Department of Moscow" Site #643009, Moscow
  - FSBI Russian Oncological Scientific Center named after N.N. Blokhina of RAMS, 23 Site #643001, Moscow
  - Federal State Budgetary Health care Institution "Central clinical hospital of Russian Academy of Science (CCH RAS), in-patient unit, urological department Site #643005, Moscow
  - FSI Moscow Research Oncological Institute named after P.A.Gertsen Site #643003, Moscow
  - Medical radiology research center named after A.F. Tsyba - branch of FSBI "National Medical Research Center of Radiology" of Ministry of healthcare of Russian Federation Site #643008, Obninsk
  - Budgetary Health care Institution of Omsk region "Clinical oncological dispensary" Site #643007, Omsk
  - SBHI Sverdlovskaya Regional Clinical Hospital #1 Site #643004, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in male subjects with high-risk prostate cancer who had undergone radical prostatectomy (RP) in 18 sites in China and Russia between Dec 2012 and Sep 2019. The study participation for each subject was at least 36 months. The end of study was when 61 biochemical relapse (BR) events were observed on the study global level.
Pre-assignment Details: Subjects had to have undergone RP no more than 8 weeks prior to randomisation, with post-RP prostate specific antigen (PSA) levels ≤0.2 nanograms/millilitre (ng/mL). The screening visit took place 6 weeks after RP (i.e. 2 weeks prior to randomisation). No other treatment for prostate cancer was permitted.
Groups:
- Active Surveillance: Subjects were treated according to each study centre's standard of care. No adjuvant treatment with any method (hormonal treatment and/or surgical castration and/or radiation therapy) was initiated prior to evidence of disease progression (clinical or biochemical).
- Triptorelin: Subjects were treated with triptorelin as a hormonal adjuvant to RP and received intramuscular injections of 11.25 milligrams (mg) triptorelin every 3 months for a total of 3 injections (at baseline, 3 months and 6 months).
Period: Overall Study
Arm/Group | Active Surveillance | Triptorelin
Started | 117 | 109
Received Triptorelin Treatment | 0 | 105
Completed (Completed study at Month 36 or completed Follow-up) | 76 | 73
Not Completed | 41 | 36
Not completed — Lost to Follow-up | 7 | 2
Not completed — Withdrawal by Subject | 26 | 23
Not completed — Adverse Event (up to Month 36) | 1 | 1
Not completed — Death | 0 | 2
Not completed — Did not attend end of study visit | 7 | 8

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population consisted of all randomised subjects analysed according to the group to which they were randomised (i.e. regardless of treatment approach followed).
Groups:
- Triptorelin: Subjects were treated with triptorelin as a hormonal adjuvant to RP and received intramuscular injections of 11.25 mg triptorelin every 3 months for a total of 3 injections (at baseline, 3 months and 6 months).
- Total: Total of all reporting groups
Arm/Group | Active Surveillance | Triptorelin | Total
Number analyzed (Participants) | 117 | 109 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (6.8) | 65.4 (6.1) | 65.3 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 117 | 109 | 226
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 84 | 79 | 163
  Caucasian / White | 33 | 30 | 63
Region of Enrollment [Count of Participants; unit: Participants]
  China | 84 | 79 | 163
  Russia | 33 | 30 | 63
PSA Levels [Median (Inter-Quartile Range); unit: ng/mL] — PSA levels were measured 6 weeks after RP at the screening visit (Day -14) and these were considered as the baseline values (i.e. no separate PSA measurement was taken at the baseline visit on Day 1).
  ng/mL | 0.074 [0.074 to 0.074] | 0.074 [0.074 to 0.074] | 0.074 [0.074 to 0.074]
Testosterone Levels [Median (Inter-Quartile Range); unit: nanograms per deciliter (ng/dL)] — Testosterone levels were evaluated on blood samples taken before triptorelin injection at baseline (Day 1). Population: Only in subjects in the triptorelin arm with data available were included in the analysis.
  nanograms per deciliter (ng/dL)
    number analyzed (Participants) | 0 | 106 | 106
    (all) |  | 462.00 [333.00 to 612.00] | 462.00 [333.00 to 612.00]
Functional Assessment of Cancer Therapy - Prostate (FACT-P) Total Score [Mean (Standard Deviation); unit: scores on a scale] — The total FACT-P score is composed of 27 general questions about physical, social, emotional, and functional well-being, as well as a 12-item questionnaire about prostate-specific concerns. The total FACT-P score was calculated as the sum of 39 item scores (range of 0-156); higher scores indicate a better quality of life (QoL). Population: Only subjects with data available were included in the analysis.
  scores on a scale
    number analyzed (Participants) | 117 | 106 | 223
    (all) | 113.26 (18.64) | 114.98 (18.31) | 114.08 (18.46)
36-Item Short Form Health Survey (SF-36) Score [Mean (Standard Deviation); unit: scores on a scale] — The SF-36 health survey contains 36 items covering 8 health domains: physical functioning (PF), role-physical, bodily pain (BP), social functioning (SF), mental health (MH), role-emotional (RE), vitality (VT) and general health (GH). Subscale scores were normed to the 2009 US general population (mean=50; standard deviation [SD]=10) to give norm-based scores. Two summary measures were then calculated: PCS was derived from PF, role-physical, BP and GH; MCS was derived from SF, MH, RE and VT. The PCS and MCS norm-based scores ranged 0-100; higher scores indicate a better QoL. Population: Only subjects with data available were included in the analysis
  scores on a scale
    Physical Component Summary (PCS): number analyzed (Participants) | 117 | 104 | 221
    Physical Component Summary (PCS) | 46.31 (6.49) | 47.37 (6.62) | 46.81 (6.56)
    Mental Component Summary (MCS): number analyzed (Participants) | 117 | 104 | 221
    Mental Component Summary (MCS) | 48.18 (9.78) | 47.41 (9.59) | 47.81 (9.67)
Gleason Score Prior to RP - Total Score in Categories [Count of Participants; unit: Participants] — The Gleason score is an indication of prognosis based on prostate pathology. The total score ranges from 2 to 10 (ie, "1+1" to "5+5") with a higher score reflecting less-differentiated tumors with worse prognosis. The total score is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5). Population: Only subjects with data available were included in the analysis.
  Participants
    number analyzed (Participants) | 111 | 105 | 216
    ≤ 6 | 31 | 27 | 58
    = 7 (3+4) | 32 | 27 | 59
    = 7 (4+3) | 19 | 20 | 39
    ≥ 8 | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With BR Events
Description: The primary efficacy analyses of Biochemical Relapse-Free Survival (BRFS) was performed after 61 BR events were observed on the study global level. The number of subjects with BR events per treatment group is reported. The definition of BR was increased PSA >0.2 ng/mL confirmed by a second measurement performed 4 to 6 weeks later.
Time Frame: Baseline (Day 1) and every 3 months until end of study with final analysis performed after required 61 BRs were observed on global study level. Minimum monitoring period of 36 months for each subject; maximum duration of 78 months (last subject censored).
Population: The ITT population consisted of all randomised subjects analysed according to the group to which they were randomised (i.e. regardless of treatment approach followed).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 109
Participants | 35 | 26

2. Primary Outcome: Median Time to BRFS
Description: BRFS was defined as the time from randomisation to time of BR. The definition of BR was increased PSA >0.2 ng/mL confirmed by a second measurement performed 4 to 6 weeks later. The time point at which the first elevated PSA measurement >0.2 ng/mL was recorded was deemed to be the time of BR. The Kaplan-Meier method was used to obtain the estimates of median and/or first quartile (Q1) (if median was not reached) time to BRFS associated with each treatment. This outcome measure reports median time to BRFS (with Q1 time to BRFS reported in the subsequent outcome measure).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 109
months | NA [NA to NA] — The median time to BRFS could not be estimated due to low numbers of events. | NA [NA to NA] — The median time to BRFS could not be estimated due to low numbers of events.
Statistical Analysis 1: Comparison: Active Surveillance vs Triptorelin; A two-sided log-rank test was used to compare time to BRFS between both treatment groups; Test type: Other; p = 0.158, Log Rank; Analysis on BRFS was based on 61 BR events (comprised of 35 BR events in the active surveillance arm and 26 BR events in the triptorelin arm)
Statistical Analysis 2: Comparison: Active Surveillance vs Triptorelin; Comparison between treatment groups: Triptorelin compared to Active surveillance. A Cox proportional hazard model was fitted to compute hazards ratios (HRs) and the corresponding 95% CIs with treatment group, country (China as reference), centre (the largest centre as reference), and Gleason score on prostatectomy specimen (in categories: ≤6 / =7 / ≥8, with ≤6 considered as the reference) as fixed factors; Test type: Other; p = 0.100, Regression, Cox; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.38 to 1.09]
Statistical Analysis 3: Comparison: Active Surveillance vs Triptorelin; Comparison between countries: Russia compared to China. A Cox proportional hazard model was fitted to compute HRs and the corresponding 95% CIs with treatment group, country (China as reference), centre (the largest centre as reference), and Gleason score on prostatectomy specimen (in categories: ≤6 / =7 / ≥8, with ≤6 considered as the reference) as fixed factors; Test type: Other; p = 0.502, Regression, Cox; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.46 to 4.79]; Interactions effect between treatment group and each covariate (country, centre(country) and Gleason score) were tested one by one in separate models. An interaction effect was considered as significant if p-value was <0.20. Interaction between treatment group and country: p=0.970
Statistical Analysis 4: Comparison: Active Surveillance vs Triptorelin; Centre effect. A Cox proportional hazard model was fitted to compute HRs and the corresponding 95% CIs with treatment group, country (China as reference), centre (the largest centre as reference), and Gleason score on prostatectomy specimen (in categories: ≤6 / =7 / ≥8, with ≤6 considered as the reference) as fixed factors; Test type: Other; p = 0.671, Regression, Cox; Interactions effect between treatment group and each covariate (country, centre(country) and Gleason score) were tested one by one in separate models. An interaction effect was considered as significant if p-value was <0.20. Interaction between treatment group and centre: p=0.241
Statistical Analysis 5: Comparison: Active Surveillance vs Triptorelin; Comparison between Gleason score categories: Gleason score of =7 compared to Gleason score ≤6. A Cox proportional hazard model was fitted to compute HRs and the corresponding 95% CIs with treatment group, country (China as reference), centre (the largest centre as reference), and Gleason score on prostatectomy specimen (in categories: ≤6 / =7 / ≥8, with ≤6 considered as the reference) as fixed factors; Test type: Other; p = 0.093, Regression, Cox; Hazard Ratio (HR) = 2.35, 95% CI 2-sided [0.87 to 6.39]; Interactions effect between treatment group and each covariate (country, centre(country) and Gleason score) were tested one by one in separate models. An interaction effect was considered as significant if p-value was <0.20. Interaction between treatment group and Gleason score: p=0.272
Statistical Analysis 6: Comparison: Active Surveillance vs Triptorelin; Comparison between Gleason score categories: Gleason score of ≥8 compared to Gleason score ≤6. A Cox proportional hazard model was fitted to compute HRs and the corresponding 95% CIs with treatment group, country (China as reference), centre (the largest centre as reference), and Gleason score on prostatectomy specimen (in categories: ≤6 / =7 / ≥8, with ≤6 considered as the reference) as fixed factors; Test type: Other; p = 0.168, Regression, Cox; Hazard Ratio (HR) = 2.03, 95% CI 2-sided [0.74 to 5.55]

3. Primary Outcome: Q1 Time to BRFS
Description: BRFS was defined as the time from randomisation to time of BR. The definition of BR was increased PSA >0.2 ng/mL confirmed by a second measurement performed 4 to 6 weeks later. The time point at which the first elevated PSA measurement >0.2 ng/mL was recorded was deemed to be the time of BR. The Kaplan-Meier method was used to obtain the estimates of median and/or Q1 (if median was not reached) time to BRFS associated with each treatment. This outcome measure reports Q1 time to BRFS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 109
months | 30.0 [18.6 to 42.1] | 39.1 [29.9 to NA] — The upper limit of 95% confidence interval (CI) could not be calculated as it was not reached.

4. Secondary Outcome: Median Time to Event-Free Survival (EFS)
Description: EFS was defined as the time from randomisation to time of first clinical disease progression or death from any cause. The Kaplan-Meier method was used to obtain the estimates of median and/or Q1 (if median was not reached) time to EFS associated with each treatment. This outcome measure reports median time to EFS (with Q1 time to EFS reported in the subsequent outcome measure).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 109
months | NA [NA to NA] — The median time to EFS could not be estimated due to low numbers of events. | NA [NA to NA] — The median time to EFS could not be estimated due to low numbers of events.
Statistical Analysis 1: Comparison: Active Surveillance vs Triptorelin; A two-sided log-rank test was used to compare time to EFS between both treatment groups; Test type: Other; p = 0.639, Log Rank; Analysis was based on 2 EFS events in the active surveillance arm and 3 EFS events in the triptorelin arm
Statistical Analysis 2: Comparison: Active Surveillance vs Triptorelin; Comparison between treatment groups: Triptorelin compared to Active surveillance. A Cox proportional hazard model was fitted to compute HRs and the corresponding 95% CIs with treatment group, country (China as reference), centre (the largest centre as reference), and Gleason score on prostatectomy specimen (in categories: ≤6 / =7 / ≥8, with ≤6 considered as the reference) as fixed factors; Test type: Other; p = 0.653, Regression, Cox; Hazard Ratio (HR) = 1.52, 95% CI 2-sided [0.24 to 9.59]
Statistical Analysis 3: Comparison: Active Surveillance vs Triptorelin; Country effect. A Cox proportional hazard model was fitted to compute HRs and the corresponding 95% CIs with treatment group, country (China as reference), centre (the largest centre as reference), and Gleason score on prostatectomy specimen (in categories: ≤6 / =7 / ≥8, with ≤6 considered as the reference) as fixed factors; Test type: Other; p = 0.999, Regression, Cox
Statistical Analysis 4: Comparison: Active Surveillance vs Triptorelin; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 1.000, Regression, Cox
Statistical Analysis 5: Comparison: Active Surveillance vs Triptorelin; Gleason score effect. A Cox proportional hazard model was fitted to compute HRs and the corresponding 95% CIs with treatment group, country (China as reference), centre (the largest centre as reference), and Gleason score on prostatectomy specimen (in categories: ≤6 / =7 / ≥8, with ≤6 considered as the reference) as fixed factors; Test type: Other; p = 0.583, Regression, Cox

5. Secondary Outcome: Q1 Time to EFS
Description: EFS was defined as the time from randomisation to time of first clinical disease progression or death from any cause. The Kaplan-Meier method was used to obtain the estimates of median and/or Q1 (if median was not reached) time to EFS associated with each treatment. This outcome measure reports Q1 time to EFS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 109
months | NA [NA to NA] — The Q1 time to EFS could not be estimated due to low numbers of events. | NA [NA to NA] — The Q1 time to EFS could not be estimated due to low numbers of events.

6. Secondary Outcome: Median Time to Overall Survival (OS)
Description: OS was defined as the time between randomisation and death from any cause. The Kaplan-Meier method was used to obtain the estimates of median and/or Q1 (if median was not reached) time to OS associated with each treatment. This outcome measure reports median time to OS (with Q1 time to OS reported in the subsequent outcome measure).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 109
months | NA [NA to NA] — The median time to OS could not be estimated due to low numbers of events. | NA [NA to NA] — The median time to OS could not be estimated due to low numbers of events.
Statistical Analysis 1: Comparison: Active Surveillance vs Triptorelin; A two-sided log-rank test was used to compare time to OS between both treatment groups; Test type: Other; p = 0.557, Log Rank; 1 death occurred in the active surveillance arm and 2 deaths occurred in the triptorelin arm

7. Secondary Outcome: Q1 Time to OS
Description: OS was defined as the time between randomisation and death from any cause. The Kaplan-Meier method was used to obtain the estimates of median and/or Q1 (if median was not reached) time to OS associated with each treatment. This outcome measure reports Q1 time to OS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 109
months | NA [NA to NA] — The Q1 time to OS could not be estimated due to low numbers of events. | NA [NA to NA] — The Q1 time to OS could not be estimated due to low numbers of events.

8. Secondary Outcome: Time to Disease-specific Mortality
Description: Disease-specific mortality was measured as the time between randomisation and death related to prostate cancer.
Time Frame: as for outcome 1
Population: Analysis was not performed for this outcome measure as no deaths due to prostate cancer were observed during the study.
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Median Time to PSA Doubling Time (PSADT)
Description: PSADT was defined as the time from the first documented PSA increase >0.2 ng/mL to the time of the first value more than twice that of the first increased value. The Kaplan-Meier method was used to obtain the estimates of median and/or Q1 (if median was not reached) PSADT associated with each treatment. This outcome measure reports median time to PSADT (with Q1 time to PSADT reported in the subsequent outcome measure).
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomised subjects analysed according to the group to which they were randomised (i.e. regardless of treatment approach followed). Only subjects with increased PSA >0.2 ng/mL and with data available were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 38 | 27
months | NA [15.2 to NA] — The median and upper limit of 95% CI could not be calculated due to low number of events. | NA [9.1 to NA] — The median and upper limit of 95% CI could not be calculated due to low number of events.
Statistical Analysis 1: Comparison: Active Surveillance vs Triptorelin; A two-sided log-rank test was used to compare PSADT between both treatment groups; Test type: Other; p = 0.525, Log Rank; Analysis was based on 9 PSADT events in the active surveillance arm and 6 PSADT events in the triptorelin arm
Statistical Analysis 2: Comparison: Active Surveillance vs Triptorelin; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.435, Regression, Cox; Hazard Ratio (HR) = 1.72, 95% CI 2-sided [0.44 to 6.73]
Statistical Analysis 3: Comparison: Active Surveillance vs Triptorelin; [analysis description as in outcome 4, analysis 3]; Test type: Other; p = 0.761, Regression, Cox
Statistical Analysis 4: Comparison: Active Surveillance vs Triptorelin; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.652, Regression, Cox
Statistical Analysis 5: Comparison: Active Surveillance vs Triptorelin; [analysis description as in outcome 4, analysis 5]; Test type: Other; p = 0.726, Regression, Cox

10. Secondary Outcome: Q1 Time to PSADT
Description: PSADT was defined as the time from the first documented PSA increase >0.2 ng/mL to the time of the first value more than twice that of the first increased value. The Kaplan-Meier method was used to obtain the estimates of median and/or Q1 (if median was not reached) PSADT associated with each treatment. This outcome measure reports Q1 time to PSADT.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 38 | 27
months | 13.4 [6.0 to NA] — The upper limit of 95% CI could not be calculated as it was not reached. | 9.1 [1.6 to NA] — The upper limit of 95% CI could not be calculated as it was not reached.

11. Secondary Outcome: Percent Change From Baseline in PSA Levels
Description: As per inclusion criterion, all subjects in both treatment groups had PSA levels ≤0.2 ng/mL at the screening visit. Starting from Month 3, any elevated PSA concentration >0.2 ng/mL had to be confirmed by a second measurement performed 4 to 6 weeks later. No confirmation test was required after evidence of disease progression (BR and/or clinical disease progression). Subjects remained in the study until Month 36, even if they had a biochemical failure (PSA levels >0.2 ng/mL); then they could enter follow-up. The percent change from baseline was defined as the percent change from the screening visit (Day -14). Percent change from baseline in PSA levels are reported as median values at Months 3, 6, 9, 12, 24 and 36. Note: the raw baseline values for PSA levels are reported in the Baseline Characteristics section.
Time Frame: Screening (Day -14) and Months 3, 6, 9, 12, 24 and 36.
Population: The ITT population consisted of all randomised subjects analysed according to the group to which they were randomised (i.e. regardless of treatment approach followed). Only subjects with data available were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 109
percent change
  Month 3: number analyzed (Participants) | 109 | 104
  Month 3 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 6: number analyzed (Participants) | 99 | 104
  Month 6 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 9: number analyzed (Participants) | 99 | 100
  Month 9 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 12: number analyzed (Participants) | 100 | 96
  Month 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 24: number analyzed (Participants) | 91 | 89
  Month 24 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 36: number analyzed (Participants) | 87 | 86
  Month 36 | 0.0 [0.0 to 25.7] | 0.0 [0.0 to 0.0]

12. Secondary Outcome: Change From Baseline in Serum Testosterone Levels
Description: Serum testosterone levels were evaluated on blood samples taken before triptorelin injection at baseline and at 3, 6 and 9 months only in subjects in the triptorelin arm. Change from baseline in testosterone levels are reported as median values at Months 3, 6 and 9. Note: the raw baseline values for testosterone levels are reported in the Baseline Characteristics section.
Time Frame: Baseline (Day 1) and Months 3, 6 and 9.
Population: The ITT population consisted of all randomised subjects analysed according to the group to which they were randomised (i.e. regardless of treatment approach followed). Only subjects in the triptorelin arm with data available were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Triptorelin
Number analyzed (Participants) | 106
ng/dL
  Month 3: number analyzed (Participants) | 101
  Month 3 | -444.60 [-599.30 to -305.20]
  Month 6: number analyzed (Participants) | 96
  Month 6 | -438.80 [-599.45 to -306.15]
  Month 9: number analyzed (Participants) | 98
  Month 9 | -429.80 [-573.90 to -304.00]

13. Secondary Outcome: Change From Baseline in FACT-P Total Score
Description: Health-Related Quality of Life (HRQoL) was assessed using the FACT-P questionnaire (v4) at baseline and at 9, 24 and 36 months. The FACT-P score is composed of 27 general questions about physical, social, emotional, and functional well-being, as well as a 12-item questionnaire about prostate-specific concerns. The total FACT-P score was calculated as the sum of 39 item scores (range of 0-156); higher scores indicate a better quality of life. Change from baseline in FACT-P total score are reported as mean values at Months 9, 24 and 36. A negative change from baseline indicates decreased QoL. Note: the raw baseline values for FACT-P total score are reported in the Baseline Characteristics section.
Time Frame: Baseline (Day 1) and Months 9, 24 and 36.
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 106
score on a scale
  Month 9: number analyzed (Participants) | 94 | 98
  Month 9 | 4.75 [0.79 to 8.70] | 0.88 [-3.04 to 4.79]
  Month 24: number analyzed (Participants) | 90 | 89
  Month 24 | 1.48 [-2.86 to 5.83] | 3.78 [0.22 to 7.33]
  Month 36: number analyzed (Participants) | 80 | 83
  Month 36 | 2.76 [-1.96 to 7.49] | 3.81 [-1.05 to 8.67]

14. Secondary Outcome: Change From Baseline in SF-36 Physical and Mental Component Summary Measures Norm-Based Scores (i.e. PCS and MCS)
Description: HRQoL was assessed using the SF-36 health survey (v2) at baseline and at 9, 24 and 36 months. The 36 items cover 8 health domains: PF, role-physical, BP, SF, MH, RE, VT and GH. Subscale scores were normed to the 2009 US general population (mean=50; SD=10) to give norm-based scores. Two summary measures were then calculated: PCS was derived from PF, role-physical, BP and GH; MCS was derived from SF, MH, RE and VT. The PCS and MCS norm-based scores ranged 0-100; higher scores indicate a better QoL. Change from baseline in SF-36 PCS and MSC norm-based scores are reported as mean values at Months 9, 24 and 36. A negative change from baseline indicates decreased QoL. Note: the raw baseline values for PCS and MSC norm-based scores are reported in the Baseline Characteristics section.
Time Frame: Baseline (Day 1) and Months 9, 24 and 36.
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance | Triptorelin
Number analyzed (Participants) | 117 | 104
score on a scale
  PCS: Month 9: number analyzed (Participants) | 94 | 96
  PCS: Month 9 | 2.78 [1.23 to 4.34] | 2.60 [1.22 to 3.98]
  PCS: Month 24: number analyzed (Participants) | 89 | 84
  PCS: Month 24 | 4.49 [2.91 to 6.06] | 3.46 [1.87 to 5.04]
  PCS: Month 36: number analyzed (Participants) | 82 | 83
  PCS: Month 36 | 4.79 [3.11 to 6.46] | 4.86 [3.15 to 6.56]
  MCS: Month 9: number analyzed (Participants) | 95 | 96
  MCS: Month 9 | 1.80 [-0.35 to 3.95] | 4.26 [2.23 to 6.28]
  MCS: Month 24: number analyzed (Participants) | 89 | 85
  MCS: Month 24 | 0.55 [-1.67 to 2.77] | 2.81 [0.69 to 4.93]
  MCS: Month 36: number analyzed (Participants) | 82 | 83
  MCS: Month 36 | 1.13 [-1.35 to 3.61] | 5.10 [2.89 to 7.31]

ADVERSE EVENTS:
Time Frame: Up to 12 months for the reporting groups 'Prior to Month 12'; up to 24 months for the reporting group 'Posterior to Month 12'. For the triptorelin arm, treatment-emergent adverse events (TEAEs) are reported. For the active surveillance arm, all adverse events (AEs) are reported (TEAEs were not applicable for this arm; all AEs were considered as non-treatment emergent since subjects did not receive any triptorelin injections).
Description: The safety population consisted of all randomised subjects who received at least 1 injection for subjects in the triptorelin arm or who underwent at least 1 day of active surveillance for subjects in the active surveillance arm. One subject randomised to the triptorelin arm continued in the study but refused all injections and was considered in the active surveillance arm for safety analysis. Note: All-cause mortality = death due to any cause; Other Adverse Events = non-serious events only.
Groups:
- Active Surveillance - Safety Population - Prior to Month 12: Representing AEs reported in the active surveillance arm from Baseline (Day 1) until prior to Month 12 (Month 12 visit excluded).
  Subjects were treated according to each study centre's standard of care. No adjuvant treatment with any method (hormonal treatment and/or surgical castration and/or radiation therapy) was initiated prior to evidence of disease progression (clinical or biochemical).
- Triptorelin - Safety Population - Prior to Month 12: Representing TEAEs reported in the triptorelin arm from Baseline (Day 1) until prior to Month 12 (Month 12 visit excluded); corresponding to 12 months after the first triptorelin injection.
  Subjects were treated with triptorelin as a hormonal adjuvant to RP and received intramuscular injections of 11.25 mg triptorelin every 3 months for a total of 3 injections (at baseline, 3 months and 6 months).
- Overall Safety Population - Posterior to Month 12: Representing AEs reported in the overall safety population from Month 12 until end of study (Month 12 up to Month 36). Since no active study drug (ie, triptorelin) was administered to any subject during this period, AEs starting from the Month 12 visit were analysed and reported overall (ie, not separately for each treatment arm).
Arm/Group | Active Surveillance - Safety Population - Prior to Month 12 | Triptorelin - Safety Population - Prior to Month 12 | Overall Safety Population - Posterior to Month 12
All-Cause Mortality (participants affected / at risk) | 1/112 | 0/105 | 2/217
Serious Adverse Events (participants affected / at risk) | 11/112 | 3/105 | 2/217
Other Adverse Events (participants affected / at risk) | 27/112 | 31/105 | 7/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Surveillance - Safety Population - Prior to Month 12 (N=112) | Triptorelin - Safety Population - Prior to Month 12 (N=105) | Overall Safety Population - Posterior to Month 12 (N=217)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneum cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Surveillance - Safety Population - Prior to Month 12 (N=112) | Triptorelin - Safety Population - Prior to Month 12 (N=105) | Overall Safety Population - Posterior to Month 12 (N=217)
Chest pain (General disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 10 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0
Platelet count decreased (Investigations) | 2 | 2 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 4 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Movement disorder (Nervous system disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 2 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2013-06-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT01753297/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT01753297/SAP_001.pdf